CLINICAL TRIAL: NCT06958328
Title: A Phase III Randomized Trial of Dose Escalated Radiation in Locally Advanced Pancreas Cancer (LAPC) Patients (LAP100)
Brief Title: Testing Higher Dose Radiation Therapy for Locally Advanced Pancreatic Cancer
Acronym: LAP100
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI011; NCI-2025-01624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GI011 (Other: NRG Oncology); NRG-GI011 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Unresectable Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; Specimen Handling; Capecitabine; Fluorouracil; dehydroftorafur; Gemcitabine; Irinotecan; irinotecan sucrosofate; Leucovorin; Magnetic Resonance Spectroscopy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Observation; Oxaliplatin; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Options 1, 2, or 3) (Active Comparator): See Detailed Description.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Gemcitabine; Drug: Irinotecan Hydrochloride; Drug: Irinotecan Sucrosofate; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Nab-paclitaxel; Other: Observation Activity; Drug: Oxaliplatin; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (dose-escalated RT) (Experimental): Patients undergo dose-escalated RT daily, every other day, or twice weekly for 5 fractions or daily for 25 fractions (with or without concurrent fluorouracil or capecitabine for 25 fractions only). The 5-fraction regimen is preferred when feasible. After completing dose-escalated RT, patients who received less than 6 months of chemotherapy at study entry are encouraged to receive the remaining chemotherapy to total 6 months of chemotherapy. Patients may continue chemotherapy treatment beyond 6 months at physician's discretion. Additionally, patients undergo blood sample collection, CT, MRI and tumor tissue biopsy throughout the study. Patients may optionally undergo PET/CT prior to treatment.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Capecitabine; Procedure: Computed Tomography; Radiation: Dose-escalated Radiation Therapy; Drug: Fluorouracil; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given capecitabine
  Other Names: Ro 09-1978/000; Xeloda
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Dose-escalated Radiation Therapy — Undergo dose-escalated radiation using intensity-modulated radiation therapy treatment planning
  Other Names: Dose-escalated RT
  Arms: Arm II (dose-escalated RT)
Drug: Fluorouracil — Given fluorouracil
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine — Given gemcitabine
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Arm I (Options 1, 2, or 3)
Drug: Irinotecan Hydrochloride — Given irinotecan hydrochloride
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
  Arms: Arm I (Options 1, 2, or 3)
Drug: Irinotecan Sucrosofate — Given liposomal irinotecan
  Other Names: inotecan Hydrochloride as Sucrosulfate Salt Form Liposomal Formulation; Irinotecan Liposome; Irinotecan Sucrosofate Liposome; Irinotecan Sucrosofate-containing Pegylated Liposomal Formulation; MM 398; MM-398; MM398; nal-IRI; Nanoliposomal Irinotecan; Nanoliposomal Irinotecan as Sucrosofate; Nanoparticle Liposome Formulation of Irinotecan; Onivyde; PEP 02; PEP-02; PEP02
  Arms: Arm I (Options 1, 2, or 3)
Drug: Leucovorin Calcium — Given leucovorin calcium
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm I (Options 1, 2, or 3)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Nab-paclitaxel — Given nab-paclitaxel
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
  Arms: Arm I (Options 1, 2, or 3)
Other: Observation Activity — Undergo observation
  Other Names: Observation
  Arms: Arm I (Options 1, 2, or 3)
Drug: Oxaliplatin — Given oxaliplatin
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
  Arms: Arm I (Options 1, 2, or 3)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo standard radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm I (Options 1, 2, or 3)

SUMMARY:
This phase III trial compares the effect of dose-escalated radiation therapy to usual care in patients with locally advanced unresectable pancreatic ductal adenocarcinoma who have received an initial 4-6 months of chemotherapy. Usual care options include additional chemotherapy, observation, or standard lower-dose radiation therapy. These treatments may delay tumor growth but have not been shown to improve survival. Radiation therapy uses high energy X-rays to kill cancer cells and shrink tumors. Dose-escalated radiation therapy involves the precise delivery of higher doses to the tumor, often over a shorter period of time. This trial assesses whether using dose-escalated radiation therapy can prolong survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether dose-escalated radiation therapy (RT) improves 3-year overall survival (OS) compared to standard treatments without dose-escalated RT, in locally advanced pancreatic cancer patients without radiographic progression and with biochemical response after an initial interval of chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate and compare local progression between the two treatment arms. II. To evaluate and compare progression-free survival (PFS) between the two treatment arms.

III. To evaluate and compare chemotherapy-free interval between the two treatment arms.

IV. To evaluate and compare toxicity within and between the two treatment arms.

HEALTH-RELATED QUALITY-OF-LIFE (HRQOL) OBJECTIVES:

I. Primary: To compare Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) Total Score at 6 months between the two treatment arms.

II. Secondary: To compare nadir of HRQoL scores over course of study participation between the two treatment arms.

III. Secondary: To evaluate HRQoL scores over time between the two treatment arms.

EXPLORATORY OBJECTIVE:

I. Biospecimen collection for future correlative analyses.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (STANDARD OF CARE): Patients are assigned to 1 of 3 treatment options per physician's decision.

OPTION 1: Patients continue to receive fluorouracil, irinotecan hydrochloride, leucovorin calcium, and oxaliplatin (FOLFIRINOX or modified FOLFIRINOX [mFOLFIRINOX]) or fluorouracil, liposomal irinotecan, leucovorin calcium, and oxaliplatin (NALIRIFOX) or gemcitabine/nab-paclitaxel per standard of care for a total of 6 months of treatment. Patients may continue treatment beyond 6 months at physician's discretion.

OPTION 2: Patients undergo standard dose radiation therapy once daily for 28 or 30 fractions and receive concurrent fluorouracil or capecitabine per standard of care during radiation therapy. After completing concurrent chemoradiation, patients who received less than 6 months of chemotherapy at study entry are encouraged to receive the remaining chemotherapy to total 6 months of chemotherapy. Patients may continue chemotherapy treatment beyond 6 months at physician's discretion.

OPTION 3: Patients undergo observation per standard of care. (It is recommended [but not required] that this option only be for patients that have already completed total 6 months chemotherapy pre-randomization.)

Additionally, patients undergo blood sample collection, computed tomography (CT), magnetic resonance imaging (MRI) and tumor tissue biopsy throughout the study. Patients may optionally undergo positron emission tomography (PET)/CT prior to treatment.

ARM II (DOSE-ESCALATED RADIATION THERAPY): Patients undergo dose-escalated RT daily, every other day, or twice weekly for 5 fractions or daily for 25 fractions (with or without concurrent fluorouracil or capecitabine for 25 fractions only). The 5-fraction regimen is preferred when feasible. After completing dose-escalated RT, patients who received less than 6 months of chemotherapy at study entry are encouraged to receive the remaining chemotherapy to total 6 months of chemotherapy. Patients may continue chemotherapy treatment beyond 6 months at physician's discretion. Additionally, patients undergo blood sample collection, CT, MRI and tumor tissue biopsy throughout the study. Patients may optionally undergo PET/CT prior to treatment.

Patients are followed every 3 months from study entry for 2 years then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* At time of enrollment, the patient must have received 4-6 months of active chemotherapy with FOLFIRINOX or NALIRIFOX or gemcitabine/nab-paclitaxel. Patients are permitted to receive more than 1 type of chemotherapy for toxicity reasons, but not for disease progression. "Active chemotherapy" refers to time on chemotherapy not counting treatment breaks (i.e. if a patient had 1 month of chemotherapy followed by 1 month break, this would count as 1 month chemotherapy). Study registration must occur within 45 days of last day of chemotherapy cycle
* BASELINE PRE-ENTRY CHEMOTHERAPY REQUIREMENTS:
* Pathologically (histologically or cytologically) proven diagnosis of pancreatic ductal adenocarcinoma
* Locally advanced unresectable disease (as defined per the National Comprehensive Cancer Network [NCCN] guidelines and institutional tumor board review)
* Patients must have baseline pre-chemotherapy scans for staging. Options include: CT chest/abdomen/pelvis, CT chest/MRI abdomen/pelvis, CT chest/CT pelvis/MRI abdomen, or PET/CT performed prior to enrollment
* Age ≥ 18 years
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Required initial laboratory values:

All laboratory values must be obtained any time prior to initiation of chemotherapy up to 30 days post initiation of chemotherapy

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
* BASELINE CA19-9 AND BILIRUBIN REQUIREMENTS: The purpose is to obtain a baseline CA19-9 in the setting of a normal (or close to normal) bilirubin, since serologic response by serial CA19-9 measurements is part of post-chemotherapy eligibility criteria

  * If baseline CA19-9 > 37 U/mL the concurrent bilirubin must be ≤ 1.5 x ULN. (Note: if the bilirubin is not ≤ 1.5 x ULN both the CA19-9 and concurrent bilirubin can be repeated until bilirubin is ≤ 1.5 x ULN, as long as done within specified timeframe [up to 30 days post chemotherapy initiation])
  * If baseline CA19-9 U/mL ≤ 37, there are no restrictions on the required concurrent bilirubin level, and this can be the accepted baseline value

    * Prior radiation treatment
* Has the patient had prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Prior non-overlapping radiation (e.g., breast, head and neck, extremity) is permitted
* If uncertain about prior overlap, please contact the study principal investigator, Dr. Nina Sanford

  * POST PRE-ENTRY CHEMOTHERAPY REQUIREMENTS:
  * If baseline CA19-9 is elevated (defined as > 37 u/mL) the post-pre-entry chemotherapy CA19-9 must be less than 37 u/mL or a 50% decline from pre-chemotherapy level with absolute value less than 100u/mL
  * If baseline CA19-9 is not elevated (defined as ≤ 37 u/mL) the post-pre-entry chemotherapy CA19-9 must remain ≤ 37 u/mL
  * No active duodenal or gastric ulcers
  * No direct tumor invasion of the bowel or stomach
  * Restaging scans showing at least stable disease (no progression). Options for scans include: CT chest/abdomen/pelvis, CT chest/MRI abdomen/pelvis, or CT chest/CT pelvis/MRI abdomen, or PET/CT performed prior to enrollment, with restaging CT showing at least stable disease
  * Not pregnant and not nursing
  * No cardiac condition that was the primary reason for hospitalization in the last 6 months
  * New York Heart Association Functional Classification II or better (NYHA Functional Classification III/IV are not eligible) (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2030-10-21 (Estimated); Study Completion 2030-10-21 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to the date of death or last follow-up, assessed up to 3 years
  OS will be estimated by the Kaplan-Meier method (Kaplan 1958). The 3-year OS estimates between the two arms will be compared using a Z-test. A logistic regression model will be used to analyze the effects of factors, in addition to treatment, including, but not limited to the stratification factor, which may be associated with 3-year OS. The primary hypothesis of improved 3-year OS will be tested with a 1-sided significance level of 0.023 (level based on not having stopped at either of the 2 planned interim analyses).

SECONDARY OUTCOMES:
Local progression (LP) | From randomization to date of failure, date of death (competing event), or last known follow-up date, assessed up to 5 years
  Defined as progression of the primary tumor/nodes as determined by Response Evaluation Criteria in Solid Tumors criteria. LP will be estimated by the cumulative incidence method (Kalbfleish 1980), with death as a competing risk, and compared between treatment arms using Gray's test (Gray 1988). The Fine-Gray regression model will be used to analyze the effects of factors, in addition to treatment, which may be associated with LP (Fine 1999).
Progression-free survival (PFS) | From the date of randomization to the date of first PFS failure or last follow-up for patients without a reported PFS event, assessed up to 5 years
  Defined as local progression, distant failure, or death due to any cause. PFS will be estimated by the Kaplan-Meier method (Kaplan 1958) and estimates between treatment arms will be compared using the log-rank test (Mantel 1966). The Cox proportional hazard regression model will be used to analyze the effects of factors, in addition to treatment, which may be associated with PFS (Cox 1972).
Chemotherapy-free interval (CFI) | From the date of last dose of initial chemotherapy to the date of first dose of second line chemotherapy for progression, assessed up to 5 years
  Defined as the time in months without chemotherapy for locally advanced pancreatic cancer post the initial chemotherapy treatment. Mean CFI will be compared between treatment arms using a Z-test. Regression modeling will be used to analyze the effects of factors, in addition to treatment, which may be associated with CFI.
Long-term radiation-related ≥ grade 3 adverse events | Up to 1 year after randomization
  The percentage of patients on the dose-escalated radiation therapy arm will be reported.
Incidence of ≥ grade 3 adverse events | Up to 90 days after randomization
  The percentage of patients will be compared between the treatment arms using a Z-test.

OTHER OUTCOMES:
Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) total score at 6 months | At 6 months
  Mean FACT-Hep total score at 6 months will be compared between treatment arms using a t-test, if normality is met, or Wilcoxon test if not. Regression modeling will be used to analyze the effects of factors (e.g. stratification factor and other relevant baseline factors), in addition to treatment, that may be associated with 6-month mean FACT-Hep Total Score.
FACT-Hep score nadir | From baseline to 24 months from randomization
  The nadir is defined as the lowest score after baseline assessment. Mean nadir (for each of total score and Hep subscale) will be compared between treatment arms using a t-test, if normality is met, or Wilcoxon test if not, using 2-sided alpha=0.01 to account for multiple comparisons.
FACT-Hep total score over time | From baseline to 24 months from randomization
  Longitudinal analyses incorporating all follow-up time points will be done using longitudinal linear modeling methods to assess FACT-Hep Total Score trends across time. Baseline scores, treatment arm, time, treatment by time interaction (if significant), the stratification factor, and relevant covariates will be included in the model analyses. Other than baseline score, treatment arm, and time, only covariates with a 2-sided p-value < 0.01, to account for multiple comparisons, will be retained in the model.

CONTACTS AND LOCATIONS:
Overall Officials: Nina N Sanford, Principal Investigator — NRG Oncology
Locations (242):
- United States (242):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Arizona Center for Cancer Care, Tempe, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin